CLINICAL TRIAL: NCT05160584
Title: A Prospective, Multinational Study of Real-Life Current Standards of Care in Patients With Relapsed and/or Refractory Multiple Myeloma
Brief Title: A Study of Real-Life Current Standards of Care in Participants With Relapsed and/or Refractory Multiple Myeloma
Acronym: MoMMent
Status: Recruiting | Type: Observational
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Other Study IDs: CR109118; 64407564MMY4001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-12-15; First posted 2021-12-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Relapsed/Refractory Multiple Myeloma: Participants with relapsed/refractory multiple myeloma (RRMM) receiving antimyeloma treatment as standard of care (SOC) under routine clinical practice will be observed. The primary data source will be medical records of each participant.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is no interventional treatment component for participants with RRMM in this study.

SUMMARY:
The purpose of this study is to assess in real-life clinical practice, over a 24-month period, the effectiveness and safety and patient-reported outcomes (PROs) associated with standard of care (SOC) antimyeloma treatments in participants with previously treated relapsed and/or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* For Period 1 and 2: Have a documented diagnosis of multiple myeloma according to International myeloma working group (IMWG) diagnostic criteria. For Period 3: Start of talquetamab for the treatment of a documented diagnosis of relapsed and/or refractory multiple myeloma (RRMM) according to IMWG diagnostic criteria and the approved indication. The decision to start talquetamab must be made independently of the decision to participate in the study, with the start of treatment occurring up to 28 days following the start of screening or having occurred up to 21 days before the informed consent form (ICF) date
* For Period 1 and 2: Have an Eastern Cooperative Oncology Group (ECOG) Performance Status grade of 0 or 1. For Period 3: Have ECOG performance status of 0,1 or 2
* For Period 1,2 and 3: Must not be pregnant or must not plan to become pregnant within the study period
* For Period 1,2 and 3: Participants must sign an ICF indicating that he or she understands the purpose and observational nature of the study and is willing to participate. Consent is to be obtained prior to the initiation of any study-related data collection
* For Period 1 and 2: Received at least 3 prior lines of therapy (induction with or without hematopoietic stem cell transplant and with or without maintenance therapy is considered a single regimen). Undergone at least 1 complete cycle of treatment for each line of therapy, unless progressive disease (PD) was the best response to the line of therapy
* For Period 1 and 2: Must have documented evidence of progressive disease based on participating physician's determination of response by the IMWG response criteria on or after the last regimen. Participants with documented evidence of progressive disease within the previous 6 months and who are refractory or non-responsive to their most recent line of treatment afterwards are also eligible
* For Period 1 and 2: Measurable disease at screening as defined by any of the following: Serum monoclonal paraprotein (M-protein) level 1.0 g/dL or urine M-protein level 200 mg/24 hours; or Light chain multiple myeloma without measurable disease in the serum or the urine: Serum immunoglobulin free light chain 10 mg/dL and abnormal serum immunoglobulin kappa lambda free light chain ratio
* Period 1: Received as part of previous therapy a PI, an IMiD, and an anti-CD38 antibody (prior exposure can be from different monotherapy or combination regimens)
* Period 2: Received as part of previous therapy a PI, an IMiD, an anti-CD38 antibody, and BCMA-targeted therapy (prior exposure can be from different monotherapy or combination regimens)
* For period 3: At least one of the following prior to the start of talquetamab: a. Measurable disease at screening as defined by any of the following: Serum monoclonal paraprotein (M-protein) level greater than or equal to (>=) 0.5 grams per deciliter (g/dL) or urine M-protein level >= 200 milligram (mg) /24 hours; or b. serum immunoglobulin free light chain >= 10 milligrams per deciliter (mg/dL) and abnormal ratio of involved and uninvolved free light chains or c. presence of bone lesions or plasmacytomas (>=1 lesion has 2 diameters >= 1 centimeter [cm])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of participants with previously treated multiple myeloma, having received standard of care (SOC) antimyeloma treatments during local clinical practices.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-11-18 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to 52 months
  Overall Response Rate is defined as the percentage of participants who achieve a partial response (PR) or better response according to the International Myeloma Working Group (IMWG) response criteria, as assessed by Response Review Committee (RRC).

SECONDARY OUTCOMES:
Very Good Partial Response (VGPR) Rate | Up to 52 months
  VGPR rate is defined as the percentage of participants who achieve a VGPR or better response according to IMWG response criteria.
Complete Response (CR) Rate | Up to 52 months
  CR rate is defined as the percentage of participants who achieve a CR or better response according to IMWG response criteria.
Stringent Complete Response (sCR) Rate | Up to 52 months
  sCR rate is defined as the percentage of participants who achieve a sCR according to IMWG response criteria.
Minimal Residual Disease (MRD) Negative Rate | Up to 52 months
  MRD negative rate is defined as the percentage of participants with negative MRD status according to IMWG response criteria.
Clinical Benefit Rate (CBR) | Up to 52 months
  CBR is defined as the percentage of participants with clinical benefit. CBR=ORR (sCR + CR + VGPR + PR) + minimal response (MR).
Duration of Response (DOR) | Up to 52 months
  DOR is defined as time from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease as defined in the IMWG criteria.
Time to Response (TTR) | Up to 52 months
  TTR is defined as the time between the date of Day 1 of Cycle 1 and the first clinical response evaluation that the participant has met all criteria for PR or better response.
Time to Best Response | Up to 52 months
  Time to best response is defined as the time between the date of Day 1 of Cycle 1 and best objective response.
Time to Next Treatment (TTNT) | Up to 52 months
  TTNT is defined as the time from diagnosis to the start of the next-line treatment.
Progression-free Survival (PFS) | Up to 52 months
  PFS is defined as the time from the date of Day 1 of Cycle 1 to the date of first documented disease progression (as defined in the IMWG response criteria) or death due to any cause, whichever occurs first.
Time to Progression on the Next Line of Subsequent Antimyeloma Therapy or Death, Whichever Occurs First (PFS2) | Up to 52 months
  PFS2 is defined as the time from the date of Day 1 of Cycle 1 to progression on the next line of subsequent antimyeloma therapy or death, whichever occurs first.
Overall Survival (OS) | Up to 52 months
  OS is the duration from the date of Day 1 of Cycle 1 to the date of the participant's death or study completion, whichever occurs first.
Change from Baseline in Health-related Quality of Life (HRQoL) (Symptoms, Functioning, and Well-being) Assessed by European Organization for Research and Treatment of Cancer Quality-of-life Questionnaire Core 30 (EORTC-QLQ-C30) Scale Score | Baseline up to 52 months
  The EORTC-QLQ-C30 Version 3 includes 30 items in 5 functional scales (physical, role, emotional, cognitive, and social), 1 global health status scale, 3 symptom scales (pain, fatigue, and nausea/vomiting), and 6 single symptom items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The responses are reported using a verbal and numeric rating scales. The item and scale scores are transformed to a 0 to 100 scale. A high scale score represents a higher response level. Thus, a high score for a functional scale represents a high/healthy level of functioning and a high score for the global health status represents high HRQoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Change from Baseline in Health-related Quality of Life (HRQoL) (Symptoms, Functioning, and Well-being) Assessed by EuroQol Five Dimension Questionnaire 5-Level (EQ-5D-5L) | Baseline up to 52 months
  The EQ-5D-5L is a generic measure of health status. The EQ-5D-5L is a 5-item questionnaire that assesses 5 domains including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression plus a visual analog scale rating "health today" with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Period 1 and 2: Change from Baseline in Health-related Quality of Life (HRQoL) (Symptoms, Functioning, and Well-being) Assessed by EORTC QLQ-IL39 | Baseline up to 52 months
  EORTC QLQ-IL39 (four single items from the EORTC QLQMY20) will be performed to assess emotional health status (feel restless or agitated, thinking about your illness, worried about dying, worried about health in the future) on scale of 1 (not at all) to 4 (very much).
Number of Participants with Adverse Events (AEs) | Up to 52 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Severity of Adverse Events as Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) | Up to 52 months
  Severity of AEs has 5 grades based on CTCAE criteria: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening consequences; Grade 5: Death related to adverse event.
Period 3: Number of Participants Reporting Oral Toxicities Using Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Up to 52 months
  PRO-CTCAE consist of 1-8 questions of common AEs experienced by people with cancer that are appropriate for self-reporting of treatment tolerability. Each symptom selected for inclusion can be rated by up to 3 attributes characterizing the presence/frequency, severity, and/or interference of the AEs. The following items were selected for inclusion for patients with multiple myeloma: nausea, vomiting, diarrhea, shortness of breath, rash, dizziness, headache, taste changes, and fatigue/tiredness/lack of energy.
Period 3: Number of Participants Reporting Oral Toxicity Symptoms Using the Epstein Taste Survey (ETS) | Up to 52 months
  The Epstein Taste Survey consists of 17 items from the full 71 item PRO instrument, specific to taste changes. Developed for use in patients with head and neck cancer.
Period 3: Percentage of Participants with Overall Response to Subsequent Therapies | Up to 52 months
  Overall Response Rate is defined as the percentage of participants who achieve a partial response (PR) or better response according to the International Myeloma Working Group (IMWG) response criteria, as assessed by Response Review Committee (RRC). Overall response for subsequent therapies, including BCMA-targeted therapies after treatment with talquetamab will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V., Belgium Clinical Trial, Study Director — Janssen Pharmaceutica N.V., Belgium
Locations (84):
- Austria (2):
  - LKH Leoben, Leoben
  - Krankenhaus der barmherzigen Schwestern, Vienna
- Belgium (5):
  - Ziekenhuis Oost-Limburg, Genk
  - UZ Leuven, Leuven
  - Chu Helora Hospital De Mons Site Kennedy, Mons
  - Vitaz, Sint-Niklaas
  - Ucl de Mont-Godinne, Yvoir
- France (5):
  - CHRU de Lille Hopital Claude Huriez, Lille
  - CHU de Montpellier Hopital Saint Eloi, Montpellier
  - CHU de Nantes hotel Dieu, Nantes
  - Centre hospitalier Lyon-Sud, Pierre-Bénite
  - Pôle IUC Oncopole CHU, Toulouse
- Germany (12):
  - Charite Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berin
  - Universitaetsklinikum Koeln, Cologne
  - Universitatsklinikum Carl Gustvav Carus Dresden an der Technischen Universitat Dresden, Dresden
  - Universitätsklinik Hamburg-Eppendorf - Orthopädische Universitätsklinik und Poliklinik, Hamburg
  - St. Barbara-Klinik Hamm GmbH, Hamm
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Staedtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - MVZ Mitte-Onkologische Schwerpunktpraxis, Leipzig
  - Universitaetsklinikum Leipzig, Leipzig
  - Klinikum der Eberhard Karls Universitaet Abt fur innere Med II Haematologie Onkologie Germany, Tübingen
  - Universitatsklinikum Wurzburg, Würzburg
  - Heinrich-Braun-Klinikum gGmbH, Zwickau
- Greece (8):
  - University Hospital of Alexandroupolis, Alexandroupoli
  - Henry Dunant Hospital Center, Athens
  - Laiko General Hospital of Athens, Athens
  - Alexandra Hospital, Athens
  - Metaxa Cancer Center Hospital Of Piraeus, Piraeus
  - General University Hospital of Patras, Rio
  - Anticancer Hospital of Thessaloniki Theageneio, Thessaloniki
  - Ahepa University General Hospital of Thessaloniki, Thessaloniki
- Italy (20):
  - U.O. Ematologia Istituto Tumori Giovanni Paolo II, Bari
  - Istituto di Ematologia Seràgnoli azienda ospedaliera univeristaria Policlinico S.Orsola-Malpighi, Bologna
  - Policlinico di Catania, Catania
  - Ospedale Civile di Civitanova Marche, Civitanova Marche
  - IRCCS Azienda Ospedaliera San Martino - IST, Genova
  - Ospedale Policlinico San Martino IRCCS, Genova
  - Ospedale Vito Fazzi, Lecce
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Universita degli Studi di Padova Azienda Ospedaliera di Pa, Padua
  - Ospedale Villa Sofia-Cervello, Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Presidio Ospedaliero Pescara, Pescara
  - Grande Ospedale Metropolitano 'Bianchi-Melacrino-Morelli' Reggio Calabria, Reggio Calabria
  - Università di Roma La Sapienza, Roma
  - Fondazione Policlinico Universitario A Gemelli IRCCS, Roma
  - Campus Bio Medico di Roma, Roma
  - Casa Sollievo Della Sofferenza IRCCS, San Giovanni Rotondo
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Ospedale Cardinale G. Panico, Tricase
  - Azienda Ulss 8 Berica- Ospedale Di Vicenza, Vicenza
- Netherlands (2):
  - VU Medisch Centrum, Amsterdam
  - UMCG, Groningen
- Portugal (3):
  - Ulstmad - Hosp. Chaves, Chaves
  - Uls Coimbra - Hosp. Univ. Coimbra, Coimbra
  - Uls Sao Joao - Hosp. Sao Joao, Porto
- Spain (16):
  - Inst. Cat. Doncologia-H Duran I Reynals, Barcelona
  - Hosp. de Cabuenes, Gijón
  - Hosp. Univ. Virgen de Las Nieves, Granada
  - Hosp. de Jerez de La Frontera, Jerez de la Frontera
  - Hosp. de Leon, León
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. Son Espases, Palma
  - Clinica Univ. de Navarra, Pamplona
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
  - Hosp. Clinico Univ. de Valencia, Valencia
  - Hosp. Univ. Dr. Peset, Valencia
  - Hosp. Clinico Univ. de Valladolid, Valladolid
  - Hosp. Univ. Miguel Servet, Zaragoza
- Switzerland (4):
  - Kantonsspital Graubunden, Chur
  - Kantonsspital Winterthur, Medizinische Onkologie, Winterthur
  - Hirslanden Klinik Hirslanden, Zurich
  - Universitatsspital Zurich, Zurich
- United Kingdom (7):
  - Southmead Hospital, Bristol
  - University College Hospital, London
  - Kings College Hospital, London
  - St Georges Hospital, London
  - Maidstone Hospital, Maidstone
  - Nottingham University Hospitals NHS Trust, Nottingham
  - The Royal Marsden NHS Trust Sutton, Surrey

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency

REFERENCES:
- [Derived] Einsele H, Moreau P, Bahlis N, Bhutani M, Vincent L, Karlin L, Perrot A, Goldschmidt H, van de Donk NWCJ, Ocio EM, Martinez Lopez J, Rodriguez-Otero P, Dytfeld D, Jakubowiak A, Schinke C, Besemer B, Anguille S, Manier S, Rasche L, Teipel R, Scheid C, Pawlyn C, Cavo M, Diels J, Ghilotti F, Lau BW, Renaud T, Orel O, Ong F, Ramos DF, Ammann E, Parekh T, Albrecht C, Weisel K, Mateos MV. Comparative Efficacy of Talquetamab vs. Real-World Physician's Choice of Treatment in Triple-Class-Exposed Relapsed/Refractory Multiple Myeloma: Updated Analyses of MonumenTAL-1 vs. LocoMMotion/MoMMent. Adv Ther. 2025 Nov 28. doi: 10.1007/s12325-025-03409-y. Online ahead of print. PMID 41313549
- [Derived] Einsele H, Moreau P, Bahlis N, Bhutani M, Vincent L, Karlin L, Perrot A, Goldschmidt H, van de Donk NWCJ, Ocio EM, Martinez-Lopez J, Rodriguez-Otero P, Dytfeld D, Diels J, Strulev V, Haddad I, Renaud T, Ammann E, Cabrieto J, Perualila N, Gan R, Zhang Y, Parekh T, Albrecht C, Weisel K, Mateos MV. Comparative Efficacy of Talquetamab vs. Current Treatments in the LocoMMotion and MoMMent Studies in Patients with Triple-Class-Exposed Relapsed/Refractory Multiple Myeloma. Adv Ther. 2024 Apr;41(4):1576-1593. doi: 10.1007/s12325-024-02797-x. Epub 2024 Feb 24. PMID 38402374
- [Derived] Moreau P, Mateos MV, Gonzalez Garcia ME, Einsele H, De Stefano V, Karlin L, Lindsey-Hill J, Besemer B, Vincent L, Kirkpatrick S, Delforge M, Perrot A, van de Donk NWCJ, Pawlyn C, Manier S, Leleu X, Martinez-Lopez J, Ghilotti F, Diels J, Morano R, Albrecht C, Strulev V, Haddad I, Pei L, Kobos R, Smit J, Slavcev M, Marshall A, Weisel K. Comparative Effectiveness of Teclistamab Versus Real-World Physician's Choice of Therapy in LocoMMotion and MoMMent in Triple-Class Exposed Relapsed/Refractory Multiple Myeloma. Adv Ther. 2024 Feb;41(2):696-715. doi: 10.1007/s12325-023-02738-0. Epub 2023 Dec 19. PMID 38110653